CLINICAL TRIAL: NCT02312037
Title: GEMTUZUMAB OZOGAMICIN (MYLOTARG (REGISTERED)) EXPANDED ACCESS PROTOCOL FOR TREATMENT OF PATIENTS IN THE UNITED STATES WITH RELAPSED/REFRACTORY ACUTE MYELOGENOUS LEUKEMIA WHO MAY BENEFIT FROM TREATMENT AND HAVE NO ACCESS TO OTHER COMPARABLE/ALTERNATIVE THERAPY
Brief Title: Expanded Access /Compassionate Use Protocol For Relapsed Or Refractory CD33 Positive AML Patients In The USA Without Access To Comparable Or Alternative Therapy
Acronym: AML
Status: No longer available | Type: Expanded Access
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1761026
Record Dates: First submitted 2014-12-04; First posted 2014-12-09 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: CD33 Positive Acute Myelogenous Leukemia
Keywords: Relapsed CD33 AML; Refractory CD33 AML; Relapsed CD33 APL; Refractory CD33 APL; Relapsed CD33 MDS; Refractory CD33 MDS
MeSH Terms: interventions — Gemtuzumab

INTERVENTIONS:
Biological: Antibody Drug Conjugate Chemotherapeutic — Three Treatment Regimens:
  1. Mylotarg <=9 mg/m2 as a single agent on Day 1 & 14 of a 28-day cycle for a total of two cycles
  2. Mylotarg in combination with a recognized anthracycline and/or nucleoside-antagonist containing regimen
  3. Mylotarg as monotherapy or in tested combinations with ATRA and/or arsenic trioxide for APL
  Other Names: Gemtuzumab ozogamicin

SUMMARY:
An expanded access/compassionate use protocol that allows access to Mylotarg for relapsed/refractory AML CD33 positive patients in the USA.

Contact: B1761026@iconplc.com

DETAILED DESCRIPTION:
Contact:

B1761026@iconplc.com

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of relapsed/refractory AML (defined as >=5% marrow blasts by morphology), including MDS, with persisting rising blasts and no other comparable or satisfactory alternative therapy available. If bone marrow has <5% blasts by morphology but the patient has evidence of relapse with extra-medullary disease progression. In select cases presenting with conversion of MRD from negative to positive, treatment with GO may be allowed where no alternative treatments are feasible.

OR

* Confirmed diagnosis of relapsed or refractory APL with persisting or rising leukemic burden (either by morphology, cytogenetic analysis or by molecular techniques), and no other comparable or satisfactory alternative therapy available.
* Documentation that malignant cells express CD33

  4) Age >=3 months

  5) Adequate non-hematologic organ function

Exclusion Criteria:

* Untreated AML and MDS or AML and MDS in complete remission.
* Patients with a known history of VOD/SOS.
* Patients with a known hypersensitivity to Mylotarg or its parts: hP67.6 antibody, calicheamicin derivatives or other ingredients.
* Participation in other studies involving investigational drug(s) (Phases 1-4) during study participation.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (140):
- United States (140):
  - University of Alabama at Birmingham/Children's of Alabama, Birmingham, Alabama
  - Alaska Oncology & Hematology, LLC, Anchorage, Alaska
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Banner Pediatric Specialists Hematology/Oncology Clinic, Mesa, Arizona
  - Cardon Children's Medical Center., Mesa, Arizona
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Children's Hospital Of Los Angeles - University Of Southern California School Of Medicine, Los Angeles, California
  - Kaiser Permanente - Oakland Medical Center, Oakland, California
  - Kaiser Permanente - Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Kaiser Permanente - Roseville, Roseville, California
  - UCSD/ Rady Children's Hospital, San Diego, California
  - Kaiser Permanente - Santa Clara, Santa Clara, California
  - c/o Thomas Ferencz, RPh, BCOP, Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Smilow Cancer Hospital at Yale-New Haven, New Haven, Connecticut
  - Yale New-Haven Hospital & Smilow Cancer Center, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale Medical Group, Trumbull, Connecticut
  - Nemours - A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - JDCH pediatric Oncology and Hematology, Hollywood, Florida
  - Joe Dimaggio Children's Hospital, Hollywood, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - Baptist Medical Center/Wolfson Children's Hospital, Jacksonville, Florida
  - Blood and Marrow Transplant Center, Orlando, Florida
  - Cancer Institute of Florida, Orlando, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Memorial Cancer Institute at Memorial Hospital West, Pembroke Pines, Florida
  - Memorial Hospital West, Pembroke Pines, Florida
  - Johns Hopkins All Children's Hospital IDS Pharmacy, St. Petersburg, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins All Children's Outpatient Care Pediatric Hematology/Oncology Department, St. Petersburg, Florida
  - H.Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - The Blood & Marrow Transplant Group Of Georgia, Atlanta, Georgia
  - Children's Healthcare of Atlanta at Scottish Rite, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Investigational Drugs Service Pharmacy, Attn. Judy Pi, PharmD, Ami Patel, PharmD, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center/Loyola University Medical Center, Maywood, Illinois
  - Loyola University Chicago, performing research at Loyola University Medical Center, Maywood, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Indiana University Riley Hospital for Children, Indianapolis, Indiana
  - IU Health Pharmacy, Indianapolis, Indiana
  - Indiana Blood and Marrow Transplantation - Administrative Offices, Indianapolis, Indiana
  - Indiana Blood and Marrow Transplantation, Indianapolis, Indiana
  - St.Francis Hospital, Indianapolis, Indiana
  - University of Kansas Hospital, Kansas City, Kansas
  - The University of Kansas Cancer Center and Medical Pavilion, Westwood, Kansas
  - The University of Kansas Cancer Center and Medical Pavillion, Westwood, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - UK Healthcare Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University IDS Pharmacy, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - The West Clinic, P.C. dba West Cancer Center, Southaven, Mississippi
  - Siteman Cancer Center - West County, Creve Coeur, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, Siteman Cancer Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center - South County, St Louis, Missouri
  - Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore Hematology Oncology Associates, P.C., East Setauket, New York
  - Weill Cornell Medical College - New York-Presbyterian Hospital, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - University of Rochester Cancer Center Pharmacy, Rochester, New York
  - University of Rochester Medical Center, Rochester, New York
  - Brody School of Medicine at ECU, Greenville, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - University Hospitals of Cleveland Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Geisinger Medical Center, Danville, Pennsylvania
  - Milton Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Thomas Jefferson University (Tju) - Jefferson University Physicians (Jup), Philadelphia, Pennsylvania
  - Thomas Jefferson University, Investigative Drug Service, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Trials Office (Clinical), Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center, Clinical Trials Office (Regulatory), Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Allegheny Health Network, Cancer Institute, West Penn Hospital, Pittsburgh, Pennsylvania
  - The West Clinic, P.C. dba West Cancer Center, Germantown, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Baptist Memorial Hospital, Memphis, Tennessee
  - The West Clinic, P.C. dba West Cancer Center, Memphis, Tennessee
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Sarah Cannon Center for Blood Cancer, Nashville, Tennessee
  - Tennessee Oncology - Nashville, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - TriStar Centennial Medical Center/Sarah Cannon Cener for Blood Cancer, Nashville, Tennessee
  - TriStar Centennial Medical Center, Nashville, Tennessee
  - TriStar Medical Group Children's Specialist, Nashville, Tennessee
  - VA Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - Vanderbilt University Medical Center - The Vanderbilt Clinic, Nashville, Tennessee
  - Children's Blood and Cancer Center, Austin, Texas
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Dell Children's Medical Center, Austin, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - Cook Children's Hematology/Oncology Center, Fort Worth, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Cook Children's Hematology/Oncology Center - Grapevine, Grapevine, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Texas Children's Hospital Attn: Investigational Pharmacy Services, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Houston Methodist Cancer Center, Houston, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
  - Huntsman Cancer Institute-University of Utah, Salt Lake City, Utah
  - Primary Children's Hospital, Salt Lake City, Utah
  - Cancer Center IDS Pharmacy Attn: Lauren Benusa, Pharm D., Charlottesville, Virginia
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - UVA Health System, Charlottesville, Virginia
  - Virginia Oncology Associates, Hampton, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Swedish Medical Center First Hill, IDS Pharmacy, Seattle, Washington
  - Seattle Children's IDS Pharmacy - Attn. Laura Winter, Seattle, Washington
  - Seattle Children's, Seattle, Washington
  - Lisa Nakatsu, RPh, Seattle, Washington
  - Fox Valley Hematology & Oncology, SC, Appleton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Fox Valley Hematology & Oncology, SC, Oshkosh, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, Wauwatosa, Wisconsin
  - Aurora Health Care, Aurora Cancer Care, West Allis, Wisconsin

REFERENCES:
- [Derived] Wang ES, Aplenc R, Chirnomas D, Dugan M, Fazal S, Iyer S, Lin TL, Nand S, Pierce KJ, Shami PJ, Vermette JJ, Abboud CN. Safety of gemtuzumab ozogamicin as monotherapy or combination therapy in an expanded-access protocol for patients with relapsed or refractory acute myeloid leukemia. Leuk Lymphoma. 2020 Aug;61(8):1965-1973. doi: 10.1080/10428194.2020.1742897. Epub 2020 May 20. PMID 32432489
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1761026&StudyName=Expanded%20Access%20/Compassionate%20Use%20Protocol%20For%20Relapsed%20Or%20Refractory%20CD33%20Positive%20AML%20Patients%20In%20The%20USA%20Without%20Access%20To%20Comparabl